CLINICAL TRIAL: NCT03722563
Title: Comparison of Total Laparoscopic Hysterectomy With Sacrocolpopexy Versus Total Laparoscopic Hysterectomy With Lateral Suspension in Patients With Pelvic Organ Prolapse: a Randomized Clinical Trial
Brief Title: Total Laparoscopic Hysterectomy With Sacrocolpopexy Versus Total Laparoscopic Hysterectomy With Lateral Suspension in Patients With Pelvic Organ Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, bekirsitkiisenlik, principal investigator, Antalya Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLHSvsTLHLS
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Pelvic Organ Prolapse
Keywords: lateral suspension; laparoscopic hysterectomy; pelvic organ prolapse; sacrocolpopexy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TLHS (Active Comparator): total laparoscopic hysterectomy with sacrocolpopexy will be performed
  Interventions: Procedure: total laparoscopic hysterectomy with sacrocolpopexy
- TLHLS (Experimental): total laparoscopic hysterectomy with lateral suspension will be performed
  Interventions: Procedure: total laparoscopic hysterectomy with lateral suspension

INTERVENTIONS:
Procedure: total laparoscopic hysterectomy with sacrocolpopexy — Surgical correction of anterior and/or apical pelvic organ prolapse by laparoscopy
  Arms: TLHS
Procedure: total laparoscopic hysterectomy with lateral suspension — Surgical correction of anterior and/or apical pelvic organ prolapse by laparoscopy
  Arms: TLHLS

SUMMARY:
This prospective randomized surgical trial is designed to compare objective and subjective outcomes of total laparoscopic hysterectomy with sacrocolpopexy versus total laparoscopic hysterectomy with lateral suspension for the treatment of pelvic organ prolapse

ELIGIBILITY:
Inclusion Criteria:

* Women with symptomatic pelvic organ prolapse stage II or higher (according to the International Continence Society Pelvic Organ Prolapse quantification system - POPQ) in anterior and/or apical (central) compartment that require surgical management

Exclusion Criteria:

* Patients that are not candidates for general anesthesia or laparoscopy
* Inability to consent
* history of hysterectomy
* history of anterior or apical pelvic organ prolapse surgery
* history of urinary incontinence surgery
* pregnancy or breast-feeding during the study period
* suspicious adnexal masses or other factors that may indicate pelvic malignancy

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Rate of objective cure | 12 months
  Recurrences of vaginal vault prolapse will be assessed as objective cure by using the pelvic organ prolapse quantification (POP-Q) system

SECONDARY OUTCOMES:
Patient Global Impression of Improvement (PGI-I) | 12 months
  Patient Global Impression of Improvement scale is global index that may be used to rate the response of a condition to a therapy.
  It is a 7-point scale where a score of 1 indicates that the patient is "very much improved," a score of 4 indicates that the patient has experienced "no change," and a score of 7 indicates that the patient is "very much worse."
International Consultation of Incontinence Questionnaire - Short Form (ICIQ-SF) | 12 months
  The questionnaire contains four items: frequency of urinary incontinence, amount of leakage, overall impact of urinary incontinence and self-diagnostic. The first item has 6 response categories (never, once a week, two or three times a week, once a day, a few times a day, always) and is scored from 0 to 5. The second item has 4 response categories (none, small amount, moderate amount, large amount) and is scored 0, 2, 4, or 6. The third item (how much urine leakage affects your daily life) has 5 response (not at all, mildly, moderately, severely, to a great extent) and is scored from 0 to 10. The first three items are scored and then summed to produce a total score, ranging from 0 to 21. The last item is a diagnostic item to assess the perceived cause of incontinence. This item is included upon the request of clinicians and is not used for scoring. A higher ICIQ-UI-SF score indicates higher frequency, severity, and lower quality of life.
International Consultation on Incontinence Questionnaire on Vaginal Symptoms (ICIQ-VS) | 12 months
  The questionnaire evaluates several pelvic floor dysfunctions including questions regarding intestinal, vaginal, sexual symptoms and quality of life impact. It includes 14 questions (dragging abdominal pain, vaginal soreness, reduced sensation around vagina, vagina too loose/lax, lump coming down in vagina, lump coming out of vagina, dry vagina, digitation for bowel opening, tight vagina, current sex life, worries about vagina affect sex life, relationship, sex life spoilt, overall impact on everyday life) and divided into three independent domains. Vaginal symptoms score varies from 0 to 53. Sexual symptoms score varies from 0 to 58. Quality of life impact score varies from 0 to 10. Usually each question has 3 to 5 possible answers; the higher the score, the most severe is the symptom or the negative quality of life impact.

CONTACTS AND LOCATIONS:
Overall Officials: Bekir Sıtkı İsenlik, MD, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Muratpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided